CLINICAL TRIAL: NCT00820989
Title: Inflammation and the Host Response to Injury (In Healthy Volunteers)
Acronym: Mono
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 0220013432; GM64351-01
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Immune System
Keywords: Healthy Immune System
MeSH Terms: interventions — Endotoxins; Lipopolysaccharides; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Time points after IV Endotoxin administration compared to baseline (immediately before Endotoxin administration).
  Interventions: Biological: Endotoxin, Lipopolysaccharide, LPS

INTERVENTIONS:
Biological: Endotoxin, Lipopolysaccharide, LPS — Clinical Center Reference Endotoxin, lot 2, sterile saline, 2 ng/kg, bolus IV administration (~5 minutes)
  Other Names: Sodium Chloride Solution

SUMMARY:
The body's immune response to injury or infection is very complex.Endotoxin is a man-made substance, which causes the body to "mimic" sickness (fever,chills, and achiness)for a few hours. This study is designed to determine whether certain proteins, genetics, or heart rate variability change affects the body's response to endotoxin.

DETAILED DESCRIPTION:
The body's immune response to injury or infection is very complex.Immune cell activity, the release of specific mediators(such as proteins, genetics(Deoxyribonucleic acid or DNA), the body's "instructions" for making proteins (Ribonucleic Acid or RNA) and heart rate variability (HRV,the intervals between heartbeats) may affect the body's clinical response to stress such as infection.Endotoxin is a man-made substance, which causes the body to "mimic" sickness (fever,chills, and achiness)for a few hours. This study is designed to determine whether any of the above (proteins,genetics,or HRV, etc.) correlate with or affect the body's response to endotoxin.This will enable the investigator to better understand the mechanisms involved in the immune response as well as potential therapeutic strategies to improve outcomes in patients.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as demonstrated by medical history,physical exam, and laboratory tests within 6 weeks of study.
* Written informed consent prior to the performance of any study related procedure.

Exclusion Criteria:

* History of cancer, rheumatoid arthritis, or immunological, renal, hepatic, endocrine, neurologic, heart disease or hypertension
* Recent history of alcohol or drug abuse
* Mental capacity limited to the extent that the subject cannot provide written informed consent or information regarding treatment-emergent adverse events and/or tolerance of study medication and/or study procedures
* Exposure to any experimental agent or procedure within 30 days of study
* Pregnancy or breast feeding
* Prior exposure to endotoxin in an experimental setting -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2000-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Physiological, Hematological, Immunological Responses | .5-24 hours after Endotoxin administration

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Corbett, MD, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Rutgers-RWJMS, New Brunswick, New Jersey, United States